CLINICAL TRIAL: NCT01784796
Title: Mindfulness Based Stress Reduction for Women at Risk for Cardiovascular Disease
Brief Title: Mindful Hearts Study: Mindfulness to Reduce Stress
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: VA Office of Research and Development (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: NRI 12-413
Record Dates: First submitted 2013-02-04; First posted 2013-02-06 (Estimated); Results first posted 2019-05-31 (Actual); Last update posted 2021-09-16 (Actual); Status verified 2021-08

CONDITIONS: Cardiovascular Disease; Psychological Stress; Stroke; Coronary Artery Disease
Keywords: cardiovascular disease; women's health; psychological stress; Veterans; stroke
MeSH Terms: conditions — Cardiovascular Diseases; Stress, Psychological; Stroke; Coronary Artery Disease | interventions — Mindfulness-Based Stress Reduction

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Mindfulness Based Stress Reduction (Experimental): 8 week Mindfulness Based Stress Reduction program
  Interventions: Behavioral: Mindfulness Based Stress Reduction
- Health education program (Active Comparator): 8 week Health Education program
  Interventions: Behavioral: Health Education Program

INTERVENTIONS:
Behavioral: Mindfulness Based Stress Reduction — 8 week Mindfulness Based Stress Reduction Program
  Other Names: MBSR
  Arms: Mindfulness Based Stress Reduction
Behavioral: Health Education Program — 8 week Health Education Program
  Other Names: Health Education
  Arms: Health education program

SUMMARY:
The purpose of this study is to determine how a stress reduction program, called Mindfulness Based Stress Reduction (MBSR), compared to a health education program, improves well being and reduces the risk of heart disease in women Veterans. Recruitment completed.

DETAILED DESCRIPTION:
Evidence demonstrates that chronic stress doubles the risk of myocardial infarction and contributes to proinflammatory processes implicated in coronary artery disease and stroke. Veterans who have experienced combat are at greater risk for cardiovascular disease (CVD) compared to noncombat Veterans and non-Veterans. However, previous research has focused primarily on male Veterans. Yet statistics reveal a startling number (81-92%) of women Veterans report at least one traumatic event sometime in their lives and women Veterans experience significant rates of prior life adversity such as sexual assault, physical violence, and combat exposure. Compelling evidence demonstrates a strong relationship between the breadth of prior life adversity, proinflammatory cytokines and stress-related inflammatory disease, such as CVD. Assisting women Veterans to reduce stress and develop coping strategies may improve psychological well-being and reduce CVD risk. Mindfulness Based Stress Reduction (MBSR) involves intensive training in mindfulness, which promotes positive adaptation to life stress. MBSR has been found to reduce symptoms of depression and improve quality of life in Veterans experiencing Post-Traumatic Stress Disorder (PTSD). Practitioners of MBSR gain increased awareness and insight into the relationship among their thoughts, emotions, and somatic reactivity which can facilitate change in conditioned patterns of emotional reaction. However, only minimal research and no randomized control trials (RCTs) have examined MBSR as an intervention for reducing CVD risk in women Veterans. Furthermore, previous studies have neither examined CVD risk objectively using a well-established CVD risk score nor measured endothelial dysfunction. Endothelial dysfunction is acknowledged to precede atherosclerosis and is a strong predictor of CVD. Furthermore, studies demonstrate that lifestyle changes, such exercise and yoga, can reverse endothelial dysfunction. However, no studies were found that considered endothelial function in relation to MBSR. Moreover, potential protective and risk factors, such as prior life adversity, social support, health behaviors, acculturation, and diurnal cortisol, posited to moderate the effect of psychological well-being and inflammation on MBSR have not been examined.

Women Veterans between the ages of 18 and 70 years who have at least one CVD risk factors (as defined by Framingham CVD Risk Scale) will be randomized into either an 8-week MBSR program or health education control program. The following specific aims will be addressed: (1) Determine the extent to which training in MBSR (1) improves psychological well-being, (2) decreases inflammatory burden, and (3) reduces cardiovascular risk in women Veterans; and (2) Evaluate protective and risk factors posited to moderate the effect of MBSR on psychological well being, inflammatory burden and cardiovascular risk in women Veterans. Age, body mass index (BMI), menstrual status, medications, and socioeconomic status (SES) will be evaluated as covariates. The proposed research is innovative in that MBSR has not been evaluated in women Veterans at risk for CVD. The investigators expect that MBSR will improve psychological well-being and reduce CVD risk with improvements sustained for at least 6 months. Given that CVD is a major cause of mortality, this research may have broader implications for reducing CVD in the general population.

Recruitment completed.

ELIGIBILITY:
Inclusion Criteria:

* Between the ages of 18
* Female Veteran
* Able to

  * write
  * read
  * speak English

Must have ONE of ANY of the following:

* BMI > 25
* Total cholesterol > 240
* Diabetes mellitus or pre-diabetic
* Systolic blood pressure> 120 and/or diagnosis of hypertension and/or taking antihypertensive medications
* Parental history of MI prior to age 60
* History of smoking

Exclusion Criteria:

* History of:

  * myocardial infarction or ischemic heart disease/angina
  * left ventricular hypertrophy
  * ischemic stroke
* pregnant
* planning on becoming pregnant during study period
* gave birth in prior 6 weeks or lactating
* immune-related disease
* use of immune-altering medications, such as:

  * glucocorticoids
* cancer
* active infection
* substance abuse
* major psychoses
* already trained in MBSR

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 164 (Actual)
Dates: Start 2013-07-01 (Actual); Primary Completion 2017-07-01 (Actual); Study Completion 2018-01-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Karen L. Saban, PhD RN, Principal Investigator — Edward Hines Jr. VA Hospital, Hines, IL
Locations (1):
- Edward Hines Jr. VA Hospital, Hines, IL, Hines, Illinois, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Levine GN, Lange RA, Bairey-Merz CN, Davidson RJ, Jamerson K, Mehta PK, Michos ED, Norris K, Ray IB, Saban KL, Shah T, Stein R, Smith SC Jr; American Heart Association Council on Clinical Cardiology; Council on Cardiovascular and Stroke Nursing; and Council on Hypertension. Meditation and Cardiovascular Risk Reduction: A Scientific Statement From the American Heart Association. J Am Heart Assoc. 2017 Sep 28;6(10):e002218. doi: 10.1161/JAHA.117.002218. PMID 28963100
- [Background] Saban KL, Mathews HL, Bryant FB, Tell D, Joyce C, DeVon HA, Witek Janusek L. Perceived discrimination is associated with the inflammatory response to acute laboratory stress in women at risk for cardiovascular disease. Brain Behav Immun. 2018 Oct;73:625-632. doi: 10.1016/j.bbi.2018.07.010. Epub 2018 Jul 17. PMID 30012518

RESULTS

PARTICIPANT FLOW:
Recruitment Details: We had powered the study for a total of 110 participants (55 in each group). To account for attrition, we planned on recruiting a total of 138 participants (69 in each group). We enrolled 164 participants and 136 of these completed baseline data.
Period: Overall Study
Arm/Group | Mindfulness Based Stress Reduction | Health Education Program
Started | 87 (These are participants who provided informed consent) | 77 (These are participants who provided informed consent)
Baseline Data Collected | 75 | 61
4 Week Data Collection | 48 | 41
8 wk Data Collection | 50 | 46
Completed (This is data collected 6 months after end of intervention) | 39 | 34
Not Completed | 48 | 43

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Mindfulness Based Stress Reduction | Health Education Program | Total
Number analyzed (Participants) | 75 | 61 | 136
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 71 | 59 | 130
  >=65 years | 4 | 2 | 6
Age, Continuous [Mean (Full Range); unit: years] | 50.83 [27 to 68] | 50.51 [24 to 77] | 50.75 [24 to 77]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 75 | 61 | 136
  Male | 0 | 0 | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 11 | 07 | 18
  Not Hispanic or Latino | 64 | 54 | 118
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 1 | 2
  Asian | 0 | 1 | 1
  Native Hawaiian or Other Pacific Islander | 1 | 1 | 2
  Black or African American | 29 | 26 | 55
  White | 42 | 30 | 72
  More than one race | 1 | 2 | 3
  Unknown or Not Reported | 1 | 0 | 1
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 75 | 61 | 136
Center for Epidemiological Studies Depression Scale [Mean (Standard Deviation); unit: units on a scale] — range from 0 to 60 with higher scores indicating greater depressive symptoms
  units on a scale | 22.78 (13.76) | 19.22 (11.67) | 21.17 (13.00)
Perceived Stress Scale [Mean (Standard Deviation); unit: units on a scale] — scores between 27 and 40 indicate high perceived stress
  units on a scale | 19.64 (8.21) | 17.50 (7.52) | 18.70 (8.00)
Quality of Life Index [Mean (Standard Deviation); unit: units on a scale] — range from 0 to 30 with higher scores indicating better quality of life
  units on a scale | 17.96 (6.29) | 19.16 (5.39) | 18.70 (6.30)

OUTCOME MEASURES:

1. Primary Outcome: Perceived Stress
Description: Psychological stress measured with the Perceived Stress Scale (PSS).
  Total scores on the PSS range from 0 to 40 with higher scores indicating higher levels of perceived stress. Scores between 0 to 13 suggest low stress, scores between 14 and 26 suggest moderate stress, and scores between 27 and 40 indicate high perceived stress.
Time Frame: 8 week
Population: Baseline data was compared to 8 week data (completion of program) for both the MBSR and HEP groups.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Mindfulness Based Stress Reduction | Health Education Program
Number analyzed (Participants) | 50 | 46
score on a scale | 15.94 (8.53) | 15.50 (7.33)

2. Primary Outcome: Depressive Symptoms
Description: Depressive symptoms were measured with the CES-D
  Total scores for the CES-D range from 0 to 60 with higher scores indicating greater depressive symptoms.
Time Frame: 8 week
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Mindfulness Based Stress Reduction | Health Education Program
Number analyzed (Participants) | 50 | 46
score on a scale | 18.38 (13.26) | 14.46 (11.03)

3. Primary Outcome: Quality of Life (QOL)
Description: Measured with Quality of Life Index-III Generic (QLI)
  Total scores for the QLI range from 0 to 30 with higher scores indicating better quality of life.
Time Frame: 8 week
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Mindfulness Based Stress Reduction | Health Education Program
Number analyzed (Participants) | 50 | 46
score on a scale | 19.77 (5.81) | 19.46 (5.00)

4. Secondary Outcome: Cardiovascular Risk
Description: Cardiovascular risk as measured by Reynolds Risk Score. The Reynolds Cardiovascular Risk score predicts the percent risk of having a heart attack, stroke or other major heart disease in the next 10 years. Scores range from 0 to 100% with higher scores representing greater risk of developing cardiovascular disease in 10 years.
Time Frame: 6 months
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Mindfulness Based Stress Reduction | Health Education Program
Number analyzed (Participants) | 39 | 34
score on a scale | 4.77 (3.16) | 5.80 (4.83)

ADVERSE EVENTS:
Time Frame: Duration of study and follow up - which was 6 months
Arm/Group | Mindfulness Based Stress Reduction | Health Education Program
All-Cause Mortality (participants affected / at risk) | 0/75 | 0/61
Serious Adverse Events (participants affected / at risk) | 0/75 | 0/61
Other Adverse Events (participants affected / at risk) | 1/75 | 0/61
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Mindfulness Based Stress Reduction (N=75) | Health Education Program (N=61)
Hospitalization (Gastrointestinal disorders) | 1 (1) | 0 (0) — Participant admitted to hospital for atypical chest pain later diagnosed as GERD.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2016-12-29): https://cdn.clinicaltrials.gov/large-docs/96/NCT01784796/Prot_SAP_000.pdf
  • Informed Consent Form (2016-12-14): https://cdn.clinicaltrials.gov/large-docs/96/NCT01784796/ICF_001.pdf